CLINICAL TRIAL: NCT04895007
Title: Comparative Evaluation of Covid-19 Vaccines Response and Progression in Different Covid-19 Vaccines Groups
Brief Title: Comparative Evaluation of Covid-19 Vaccines Response
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Prof.Dr.Taha Bekci, Head of Pulmonary Medicine, Karamanoğlu Mehmetbey University
Other Study IDs: 2021-04-30T1
Record Dates: First submitted 2021-05-14; First posted 2021-05-20 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: COVID-19 Vaccines
MeSH Terms: interventions — mRNA Vaccines

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group, vaccinated with Inactive Vaccine (Sinovac Life Sciences, Beijing, China).: - Any person, male or female, over 18 years of age, were vaccinated with Inactive Vaccine.
  Interventions: Biological: Covid-19 Inactive Vaccine, recombinant human adenovirus serotype number 26, mRNA VAccine
- Group, vaccinated with recombinant human adenovirus serotype number 26 (rAd26 of Sputnik V).: - Any person, male or female, over 18 years of age, were vaccinated with recombinant human adenovirus serotype number 26.
  Interventions: Biological: Covid-19 Inactive Vaccine, recombinant human adenovirus serotype number 26, mRNA VAccine
- Group, vaccinated with mRNA Vaccine (Pfizer/BionTEC).: - Any person, male or female, over 18 years of age, were vaccinated with mRNA Vaccine.
  Interventions: Biological: Covid-19 Inactive Vaccine, recombinant human adenovirus serotype number 26, mRNA VAccine

INTERVENTIONS:
Biological: Covid-19 Inactive Vaccine, recombinant human adenovirus serotype number 26, mRNA VAccine — Anti-SARS-CoV-2 IgG Antibody and Neutralizing Antibody will be evaluated 2, 6, 12 Months after second dose.

SUMMARY:
Study Population

Population with vaccinated with three different Covid Vaccines (Inactive Vaccine (Sinovac Life Sciences, Beijing, China), recombinant human adenovirus serotype number 26 (rAd26 of Sputnik V), mRNA Vaccine (Pfizer/BionTEC). This is multi center study, 5 centers will be joined to study from different part of the country. Approximately 1500 people will be enrolled to study.

DETAILED DESCRIPTION:
Aim of Study

* to evaluate Anti-SARS-CoV-2 IgG Antibody and Neutralizing Antibody response in different Vaccine Groups
* to evaluate progression of the vaccine response after 2, 6, and 12 Months after Vaccination in different Vaccine Groups, and compare antibody response in different Vaccines Group.
* It was also aimed to evaluate effect of the age, gender, co-morbid conditions such as COPD, DM, Heart Failure, Covid Infection on IgG Antibody and Neutralizing Antibody response.

Anti SARS CoV2 IgG antibody levels will be measured with chemiluminescence method (CHEM) by using ADVIA Centaur XP Immunassay System (Siemens Helthcare, GmbH, Germany) and Anti SARS CoV2 IgG reactive (Siemens Helthineers, GmbH, Germany).

Neutralizing Capacity of Anti-SARS-CoV-2 Antibodies against SARS CoV2 levels will be determined with ELISA method (ELx 808, ELISA Microplate Absorbance Reader, BioTek Instruments Inc, Winooski, VT, USA) by using Euroimmun SARS-CoV-2 NeutraLISA Assay (EUROIMMUN, Medizinische Labordiagnostika AG, Germany).

ELIGIBILITY:
Inclusion Criteria:

- Any person, male or female, over 18 years of age.

1. The patient has signed an informed consent form.
2. The patient was vaccinated with SARS-CoV-2 vaccine.

Exclusion Criteria:

* Inability to give clear information (person in an emergency, difficulty understanding the subject, etc.)
* Person under safeguard of justice
* Person under guardianship or curator ship.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: - Any person, male or female, over 18 years of age.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Anti-SARS-CoV-2 IgG Antibody and Neutralizing Antibody at 12 months | 12 Months
  * Baseline Anti-SARS-CoV-2 IgG Antibody and Neutralizing Antibody levels at 14th day after second dose
  * Change of Anti-SARS-CoV-2 IgG Antibody and Neutralizing Antibody levels at 3 Months after second dose
  * Change of Anti-SARS-CoV-2 IgG Antibody and Neutralizing Antibody levels at 6 Months after second dose
  * Change of Anti-SARS-CoV-2 IgG Antibody and Neutralizing Antibody levels at 12 Months after second dose

CONTACTS AND LOCATIONS:
Locations (4):
- Turkey (Türkiye) (4):
  - Karamanoglu Mehmetbey University, Karaman
  - Selcuk University, Konya
  - Tekirdag Namık Kemal University, Faculty of Medicine, Tekirdağ
  - Karadeniz Technic University, Faculty of Medicine, Trabzon

IPD SHARING:
Plan to Share IPD: No